CLINICAL TRIAL: NCT06358261
Title: Pilot Study of a Diabetes Prevention Patient Activation Clinical Decision Support Tool
Brief Title: Study of a Diabetes Prevention Patient Activation Clinical Decision Support Tool
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00433279; R03DK135898 (NIH)
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: PreDiabetes; Lifestyle, Healthy; Activation, Patient
MeSH Terms: conditions — Prediabetic State; Patient Participation

STUDY DESIGN:
Intervention Model Description: pilot group-randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (DPACT) (Active Comparator): In this arm, patients will have at least 2 visits with the participants primary care doctor. Before each visit, participants will complete a patient activation survey. Results of the survey will be shared with the primary care doctor and entered into the medical record so that the Diabetes Prevention Patient Activation Clinical Decision Support Tool can be used by the participants doctor during the visit to discuss lifestyle management.
  Interventions: Behavioral: Diabetes Prevention Patient Activation Clinical Decision Support Tool
- Control Arm (Usual Care) (No Intervention): Patients in the control arm will follow the same visit schedule as the intervention arm. At the beginning of the study, participants will receive a handout on pre-diabetes which will include information on lifestyle changes and the benefits of joining a Diabetes Prevention Program. Before each visit, participants will complete a patient activation survey but the results will not be shared with the participants primary care doctor

INTERVENTIONS:
Behavioral: Diabetes Prevention Patient Activation Clinical Decision Support Tool — Diabetes Prevention Patient Activation Clinical Decision Support Tool will be used by the doctor during the visit to discuss lifestyle management
  Arms: Intervention Arm (DPACT)

SUMMARY:
The investigators overarching goal is to increase the percentage of patients engaging in diabetes prevention activities to reduce the incidence of diabetes. The investigators objective is to design and pilot test a prediabetes clinical decision support (CDS) tool in the electronic health record (EHR) that will assess the patient's activation level based on responses to a questionnaire. Based on the patient's assessed level of activation, the tool will generate several communication recommendations to guide clinicians in conversations related to prediabetes/lifestyle change and tailor recommendations about available resources (e.g., care manager, health coach, DPP) to support patient activation.

DETAILED DESCRIPTION:
Patient activation, which incorporates elements of self-efficacy and readiness to change, is particularly important in managing conditions like pre-diabetes, where the mainstay of treatment is behavioral lifestyle change and self-management. Unfortunately, Primary Care Physicians (PCPs) often do not have adequate training on how to promote patient activation. Traditionally, patient decision aids are used in shared decision-making to help elicit patient preferences and guide treatment options. However, the guides primarily focus on reviewing treatment options rather than increasing patient activation, which is key to successful and efficient behavioral counseling. The Patient Activation Measure (PAM) is a widely used and validated patient-reported outcome measure for assessing patient activation. Studies have demonstrated that using PAM to tailor care to a patient's activation level decreased health service utilization while improving clinical outcomes like blood pressure and self-management behaviors.

The investigators overarching goal is to increase the percentage of patients engaging in diabetes prevention activities to reduce the incidence of diabetes. The investigators objective is to design and pilot test a pre-diabetes clinical decision support (CDS) tool in the electronic health record (EHR) that will assess the patient's activation level based on responses to a questionnaire. Based on the patient's assessed level of activation, the tool will generate several communication recommendations to guide clinicians in conversations related to pre-diabetes/lifestyle change and tailor recommendations about available resources (e.g., care manager, health coach, DPP) to support patient activation.

ELIGIBILITY:
Inclusion Criteria:

* prediabetes
* patient at Johns Hopkins General Internal Medicine clinic at Green Spring Station
* MyChart account

Exclusion Criteria:

* history of diabetes
* non-English speaker
* severe intellectual disability or psychiatric comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
patient activation as assessed by the Patient Activation Measure Survey (PAM) | baseline, 6 months
  measured by Patient Activation Measure (PAM) survey, a 13-item scale with 4 Likert response,s and scores ranging from 0 to 100 (higher score means higher activation level)

SECONDARY OUTCOMES:
number of participants referred to Diabetes Prevention Program | baseline, 6 months
  measured using electronic health record data
number of participants prescribed metformin | baseline, 6 months
  measured using electronic health record data
percent of participants who make diet changes | baseline, 6 months
  measured using survey developed by study team will assess what diet changes participants have made
change in amount and frequency of physical activity | baseline, 6 months
  measured using survey developed by study team will assess the change in amount and frequency of physical activity that participants have made

CONTACTS AND LOCATIONS:
Overall Officials: Eva Tseng, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Internal Medicine at Green Spring Station, Lutherville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No